CLINICAL TRIAL: NCT01744912
Title: A Phase I/II Study of Ublituximab in Combination With Lenalidomide (Revlimid®) in Patients With B-Cell Lymphoid Malignancies Who Have Relapsed or Are Refractory After CD20 Directed Antibody Therapy
Brief Title: Ublituximab in Combination With Lenalidomide in Patients With B-Cell Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGTX 1101-102
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Non-Hodgkins Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; B-cell Lymphomas; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Waldenstrom's Macroglobulinemia
Keywords: Lymphoma; monoclonal antibody; immunomodulatory agent; ublituximab; lenalidomide
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Lymphoma | interventions — ublituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ublituximab + Lenalidomide (Experimental): 4 cohorts, with 3 - 6 patients per cohort, as follows:
  Cohort 1: Ublituximab 450 mg + Lenalidomide 10 mg Cohort 2: Ublituximab 450 mg + Lenalidomide 15 mg Cohort 3: Ublituximab 600 mg + Lenalidomide 10 mg (escalation to 15 mg permitted after cycle 1) Cohort 4: Ublituximab 900 mg + Lenalidomide 10 mg (escalation to 15 mg permitted after cycle 1) Ublituximab is an IV infusion on days 1, 8, and 15 of cycles 1 & 2 followed by a planned maintenance with a single infusion on day 1 of cycles 3 thru 6.
  Lenalidomide is taken orally on days 9 - 28 of cycle 1 followed by daily administration on Days 1 - 28 for cycles 2 thru 6. Non-hodgkins lymphoma patients may have up to a 7 day rest period (Days 21-28) in any cycle.
  Interventions: Drug: Ublituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ublituximab — Ublituximab is a novel monoclonal antibody targeting CD20
  Other Names: TG-1101
Drug: Lenalidomide — Lenalidomide has both immunomodulatory and anti-angiogenic properties which could confer antitumor and antimetastatic effects
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine whether ublituximab in combination with lenalidomide (Revlimid®) is safe and effective in patients with B-Cell Lymphoid Malignancies who have relapsed or are refractory after CD20 directed antibody therapy.

DETAILED DESCRIPTION:
The study was intended to be a Phase 1/2 study, however, the study was terminated early and the phase 2 portion was never initiated. A limited number of participants were enrolled in Phase 1 and no maximum tolerated dose (MTD) or Phase 2 dose was identified for the combination of ublituximab and lenalidomide. Thus, Phase 2 data and results are not available to be reported.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-cell non-Hodgkins Lymphoma (NHL), Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
* Participants must have received at least one prior line of therapy with an anti-CD20 antibody (i.e. rituximab, ofatumumab, etc.) or an anti-CD20 antibody containing regimen
* Measurable or evaluable Disease
* Eastern Cooperative Oncology Group performance status 0, 1 or 2
* Participants ineligible for high dose or combination chemotherapy + stem cell transplant
* No active or chronic infection of Hepatitis B or C and no history of HIV based on negative serology
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®

Exclusion Criteria:

* Prior chemotherapy, investigational therapy or radiotherapy within 3 weeks of study entry
* Prior autologous or allogeneic stem cell transplantation within 6 months of study entry
* History of severe hypersensitivity or anaphylaxis to prior murine or mouse/human chimeric antibodies, or to any component of ublituximab, or with prior lenalidomide or thalidomide
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* History of deep vein thrombosis (DVT) or pulmonary embolus (PE) in the six months prior to Day 1 of Cycle 1
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2014-02-07 (Actual); Study Completion 2014-02-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose acceptable for participants | 4 weeks
  The Maximum Tolerated Dose will be determined by a Data Safety Monitoring Board

SECONDARY OUTCOMES:
Efficacy | After 8 weeks and then every 12 weeks
  Efficacy will include overall response rate and duration of response

OTHER OUTCOMES:
Pharmacokinetic profile including Peak Plasma Concentration (Cmax) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: TG Therapeutics Clinical Trials, Study Director — TG Therapeutics, Inc.
Locations (2):
- United States (2):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No